CLINICAL TRIAL: NCT05537948
Title: Efficacy and Safety of Pitavastatin and PCSK9 Inhibitors in Liver Transplant Patients
Acronym: PINTL
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2.0_17.03.22
Record Dates: First submitted 2022-07-01; First posted 2022-09-13 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Dyslipidemias; Hyperlipidemias; Liver Transplant Disorder; Immunosuppression; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Statins
Keywords: Dyslipidemias; Hyperlipidemias; Liver Transplant Disorder; Immunosuppression; Immunosuppressive therapy; Hydroxymethylglutaryl-CoA Reductase Inhibitors; pitavastatin; statins; PCSK9; PCSK9 Inhibitors; evolocumab; alirocumab
MeSH Terms: conditions — Dyslipidemias; Hyperlipidemias | interventions — pitavastatin

STUDY DESIGN:
Intervention Model Description: phase 1: randomized, prospective, single-center, parallel-group study
  phase 2: observational study
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- pitavastatin (Active Comparator): Pitavastatin 2 mg/d - 4 mg/d
  Interventions: Drug: Pitavastatin
- PCSK9 Inhibitors (Active Comparator): Evolocumab 140 mg once per 2 weeks or Alirokumab 150 mg once per 2 weeks
  Interventions: Drug: PCSK9 inhibitor

INTERVENTIONS:
Drug: Pitavastatin — First phase (6 months):
  Patients will be randomized 1:1 into 2 groups:
  1. pitavastatin monotherapy
  2. monotherapy with a PCSK9 inhibitor (evolocumab 140 mg or alirocumab 150 mg once every 2 weeks subcutaneously)
  In the group of Pitavastatin: Pitavastatin at visit 0 will be prescribed at a dose of 2 mg, after 1 month in the absence of side effects against the background of ongoing therapy, the dose will be increased to 4 mg.
  The lipid profile and safety of the therapy will be assessed in 1, 3 and 6 months after the start of the therapy.
  When triglyceride levels rise above 5.7 mmol/l in two consecutive analyzes, the addition of fenofibrate may be considered.
  Second phase (6 months):
  If the target level of LDL-C is not achieved during monotherapy with pitavastatin, the patient will be asked to continue treatment with combined lipid-lowering therapy (pitavastatin + PCSK9 inhibitor). There will be visits on the 7th, 9th and 12th months.
  Arms: pitavastatin
Drug: PCSK9 inhibitor — First phase (6 months):
  Patients will be randomized 1:1 into 2 groups:
  1. pitavastatin monotherapy
  2. monotherapy with a PCSK9 inhibitor (evolocumab 140 mg or alirocumab 150 mg once every 2 weeks subcutaneously)
  In the group of PCSK9 inhibitors:The lipid profile and safety of the therapy will be assessed in 1, 3 and 6 months after the start of the therapy.
  When triglyceride levels rise above 5.7 mmol/l in two consecutive analyzes, the addition of fenofibrate may be considered.
  Second phase (6 months):
  If the target level of LDL-C is not achieved during monotherapy with a PCSK9 inhibitor, the patient will be asked to continue treatment with combined lipid-lowering therapy (pitavastatin + PCSK9 inhibitor). Pitavastatin will initially be prescribed at a dose of 2 mg, after 1 month. in the absence of side effects against the background of ongoing therapy, the dose will be increased to 4 mg. There will be visits on the 7th, 9th and 12th months.
  Arms: PCSK9 Inhibitors

SUMMARY:
To study the efficacy and safety of pitavastatin and PCSK9 inhibitors in liver transplant patients on ongoing immunosuppressive therapy.

DETAILED DESCRIPTION:
1. Evaluate the efficacy and safety of lipid-lowering therapy in real clinical practice.
2. To evaluate the efficacy and safety of pitavastatin in patients undergoing liver transplantation and receiving immunosuppressive therapy.
3. Evaluate the efficacy and safety of PCSK9 inhibitors in patients undergoing liver transplantation and receiving immunosuppressive therapy.
4. To compare the efficacy and safety of pitavastatin and a PCSK9 inhibitor in patients undergoing liver transplantation and receiving immunosuppressive therapy.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent to participate in the study;
* a history of liver transplantation for any reason;
* immunosuppressive therapy;
* the presence of hyperlipidemia, requiring the prescription of lipid-lowering therapy according to the clinical guidelines of the European Society for the Study of Atherosclerosis (EAS) 2019
* failure to achieve the target level of LDL-C against the background of current lipid-lowering therapy;
* if the patient within 1 month before randomization took lipid-lowering therapy, then the absence of side effects against the background of previous lipid-lowering therapy.

Exclusion Criteria:

* treatment with PCSK9 in previous 6 months;
* current treatment in the form of lipoprotein apheresis;
* heart failure IV NYHA;
* active infectious disease, severe hematological, metabolic, gastrointestinal or endocrine dysfunctions (for example, uncontrolled thyroid dysfunction) at the time of the screening or randomization visits;
* the presence of an oncological disease, with the exception of hepatocellular carcinoma, which served as the reason for liver transplantation;
* CFR<15ml/min/1,73m2;
* pregnancy and breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
absolute change in LDL-C from baseline by months 1 and 3 of study therapy | months 1 and 3 of study therapy
  absolute change in LDL-C from baseline
percent change in LDL-C from baseline at months 1 and 3 of study therapy | months 1 and 3 of study therapy
  percent change in LDL-C from baseline
the proportion of patients who have reached the target level of LDL-C by month 1 of study therapy | month 1 of study therapy
  the proportion of patients who have reached the target level of LDL-C
the proportion of patients who have reached the target level of LDL-C by month 3 of study therapy | month 3 of study therapy
  the proportion of patients who have reached the target level of LDL-C

SECONDARY OUTCOMES:
the timing of achieving the target level of LDL-C at months 1, 3, 6, 7, 9, 12 of study therapy | months 1, 3, 6, 7, 9, 12 of study therapy
  the timing of achieving the target level of LDL-C
percent of patients with target level of LDL-C at months 6 and 12 of study therapy | months 6 and 12 of study therapy
  percent of patients with target level of LDL-C

OTHER OUTCOMES:
the proportion of patients with increased level of creatine phosphokinase (more than 4 times of the upper limit normal (ULN)) at months 1, 3, 6, 7, 9, 12 of study therapy | months 1, 3, 6, 7, 9, 12 of study therapy
  the proportion of patients with increased level of creatine phosphokinase (more than 4 times of the upper limit normal (ULN))
the proportion of patients with increase higer than the upper limit normal (ULN) of one of the parameters in blood: ALT, AST, GGT, alkaline phosphatase, total bilirubin at months 1, 3, 6, 7, 9, 12 of study therapy | months 1, 3, 6, 7, 9, 12 of study therapy
  the proportion of patients with increase higer than the upper limit normal (ULN) of one of the parameters in blood: ALT, AST, GGT, alkaline phosphatase, total bilirubin

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Ershova, PhD, Study Chair — National Medical Research Centre for Therapy and Preventive Medicine Ministry of Health of Russia
Locations (1):
- National Medical Research Centre for Therapy and Preventive Medicine of the Ministry of Health of Russia, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No